CLINICAL TRIAL: NCT00274573
Title: Acute and Long-term Effects of Once Daily Oral Inhalation of Tiotropium 18 Mcg Dry Powder Inhalation Capsules in a Placebo Controlled Parallel Group Design Study in Patients With Chronic Obstructive Pulmonary Disease (COPD) of Different Severity
Brief Title: Effects of Once Daily Tiotropium in Patients With Chronic Obstructive Pulmonary Disease (COPD) of Different Severity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.257
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium bromide

SUMMARY:
The primary objective of this study is to investigate the effect of tiotropium vs. placebo on trough FEV1 and FEV1 2 hours post inhalation after 12 weeks of treatment. For both endpoints changes from baseline will be analysed. Three strata of patients will be included (severe COPD, i.e. <35% of predicted FEV1, moderate COPD, i.e. 35% - <50% of predicted FEV1, mild COPD, i.e. 50% - 70% of predicted FEV1, according to American Thoracic Society [ATS] criteria). The study is conducted in order to find out for which endpoint tiotropium is different from placebo in which stratum.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   * Patients must have relatively stable, mild to severe airway obstruction with an FEV1 =<70% of predicted normal and an FEV1/FVC < 70 %.
   * Predicted normal values will be taken from the print-outs of the spirometers. Spirometers have to calibrated according to ECCS.
2. Male or female patients 40 years of age or older.
3. Patients must be current or ex-smokers with a smoking history of 10 or more than 10 pack-years. Pack Years = Number of cigarettes/day : 20 x years of smoking (Patients who have never smoked cigarettes must not be included)
4. Patients must be able to perform all study related tests, acceptable pulmonary function tests, including Peak Expiratory Flow Rate (PEFR) measurements, and must be able to maintain diary cards during the study period as required in the protocol.
5. Patients must be able to inhale medication from the HandiHaler.
6. All patients must sign an Informed Consent Form prior to participation in the trial i.e. prior to pre-study washout of their usual pulmonary medications.

Exclusion Criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with a recent history (i.e., one year or less) of myocardial infarction.
3. Patients with any cardiac arrhythmia requiring drug therapy or who have been hospitalised for heart failure within the past three years.
4. Patients who regularly use daytime oxygen therapy for more than 1 hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy.
5. Patients with known active tuberculosis.
6. Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed.
7. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
8. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion 1.
9. Patients with any respiratory infection in the past six weeks prior to the Screening Visit (Visit 1) or during the run-in period.
10. Patients who are currently in a pulmonary rehabilitation programme or who have completed a pulmonary rehabilitation programme in the six week prior to the Screening Visit (Visit 1).
11. Patients with known hypersensitivity to anticholinergic drugs, lactose or any other components of the inhalation capsule delivery system.
12. Patients with known symptomatic prostate hypertrophy or bladder neck obstruction.
13. Patients with known narrow-angle glaucoma.
14. Patients using oral corticosteroid medication at unstable doses (i.e., less than four weeks on a stable dose before Visit 1) or at doses in excess of the equivalent of 10 mg of prednisolone per day or 20 mg every other day.
15. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e. oral contraceptives, intrauterine devices, diaphragm or subdermal implants).
16. Patients with a history of asthma, allergic rhinitis or atopy.
17. Patients with a history of and/or active significant alcohol or drug abuse.
18. Patients who have taken an investigational drug within one month prior to Screening Visit (Visit 1). A log of all subjects screened, and reasons for exclusion for those not randomised will be maintained.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1639 (Actual)
Dates: Start 2002-03; Primary Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in trough FEV1 (Forced expiratory volume in one second) | after 12 weeks
Change from baseline in FEV1 2 hours post inhalation | after 12 weeks

SECONDARY OUTCOMES:
Change from baseline in FEV1 2 hours post inhalation | Day 1
Change from baseline in FVC (Forced Vital Capacity) 2 hours post inhalation | Day 1 and 85
Change from baseline in IVC (Inspiratory Vital Capacity) 2 hours post inhalation | Day 1 and 85
Number of patients having a COPD exacerbation | 12 weeks
Number of patients being hospitalised due to a COPD exacerbation | 12 weeks
Number of COPD exacerbations per patient | 12 weeks
Number hospitalisations due to COPD exacerbations per patient | 12 weeks
Duration of COPD exacerbations per patient | 12 weeks
Duration of hospitalisations due to a COPD exacerbation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim KG
Locations (177):
- Germany (177):
  - Boehringer Ingelheim Investigational Site, Aachen
  - Boehringer Ingelheim Investigational Site, Ahrensburg
  - Boehringer Ingelheim Investigational Site, Altenburg
  - Boehringer Ingelheim Investigational Site, Amberg
  - Boehringer Ingelheim Investigational Site, Aschaffenburg
  - Boehringer Ingelheim Investigational Site, Aue
  - Boehringer Ingelheim Investigational Site, Auerbach
  - Boehringer Ingelheim Investigational Site, Augsburg
  - Boehringer Ingelheim Investigational Site, Backnang
  - Boehringer Ingelheim Investigational Site, Bad Kissingen
  - Boehringer Ingelheim Investigational Site, Bad Krozingen
  - Boehringer Ingelheim Investigational Site, Bad Lippspringe
  - Boehringer Ingelheim Investigational Site, Bad Nauheim
  - Boehringer Ingelheim Investigational Site, Bad Neustadt an der Saale
  - Boehringer Ingelheim Investigational Site, Bad Soden
  - Boehringer Ingelheim Investigational Site, Baunatal
  - Boehringer Ingelheim Investigational Site, Beckum
  - Boehringer Ingelheim Investigational Site, Bensheim
  - Boehringer Ingelheim Investigational Site, Berlin
  - MEDARS GmbH, Berlin
  - Boehringer Ingelheim Investigational Site, Bernau
  - Boehringer Ingelheim Investigational Site, Bielefeld
  - Boehringer Ingelheim Investigational Site, Bochum
  - Boehringer Ingelheim Investigational Site, Bonn
  - Boehringer Ingelheim Investigational Site, Brake
  - Boehringer Ingelheim Investigational Site, Brandenburg
  - Boehringer Ingelheim Investigational Site, Braunschweig
  - Boehringer Ingelheim Investigational Site, Bruchsal
  - Boehringer Ingelheim Investigational Site, Buchholz
  - Boehringer Ingelheim Investigational Site, Celle
  - Boehringer Ingelheim Investigational Site, Chemnitz
  - Boehringer Ingelheim Investigational Site, Cloppenburg
  - Boehringer Ingelheim Investigational Site, Coburg
  - Boehringer Ingelheim Investigational Site, Cologne
  - Boehringer Ingelheim Investigational Site, Dachau
  - Boehringer Ingelheim Investigational Site, Darmstadt
  - Boehringer Ingelheim Investigational Site, Deggendorf
  - Boehringer Ingelheim Investigational Site, Delmenhorst
  - Boehringer Ingelheim Investigational Site, Detmold
  - Boehringer Ingelheim Investigational Site, Dillingen
  - Boehringer Ingelheim Investigational Site, Dinslaken
  - Boehringer Ingelheim Investigational Site, Dortmund
  - Boehringer Ingelheim Investigational Site, Dresden
  - Boehringer Ingelheim Investigational Site, Duisburg
  - Boehringer Ingelheim Investigational Site, Dülmen
  - Boehringer Ingelheim Investigational Site, Düren
  - Boehringer Ingelheim Investigational Site, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Eggenfelden
  - Boehringer Ingelheim Investigational Site, Eisenach
  - Boehringer Ingelheim Investigational Site, Eisenhüttenstadt
  - Boehringer Ingelheim Investigational Site, Emden
  - Boehringer Ingelheim Investigational Site, Erfurt
  - Boehringer Ingelheim Investigational Site, Erlangen
  - Boehringer Ingelheim Investigational Site, Essen
  - Boehringer Ingelheim Investigational Site, Euskirchen
  - Boehringer Ingelheim Investigational Site, Fellbach
  - Boehringer Ingelheim Investigational Site, Fluda
  - Boehringer Ingelheim Investigational Site, Frankenthal
  - Boehringer Ingelheim Investigational Site, Frankfurt
  - Boehringer Ingelheim Investigational Site, Frankfurt (Oder)
  - Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site, Freising
  - Boehringer Ingelheim Investigational Site, Fulda
  - Boehringer Ingelheim Investigational Site, Fürstenfeldbruck
  - Boehringer Ingelheim Investigational Site, Fürstenwalde
  - Boehringer Ingelheim Investigational Site, Fürth
  - Boehringer Ingelheim Investigational Site, Garmisch-Partenkirchen
  - Boehringer Ingelheim Investigational Site, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site, Germering
  - Boehringer Ingelheim Investigational Site, Goch
  - Boehringer Ingelheim Investigational Site, Göppingen
  - Boehringer Ingelheim Investigational Site, Greiz
  - Boehringer Ingelheim Investigational Site, Groß Gaglow
  - Boehringer Ingelheim Investigational Site, Großenhain
  - Boehringer Ingelheim Investigational Site, Gütersloh
  - Boehringer Ingelheim Investigational Site, Hagen
  - Boehringer Ingelheim Investigational Site, Hamburg
  - Boehringer Ingelheim Investigational Site, Hamm
  - Boehringer Ingelheim Investigational Site, Hanover
  - Boehringer Ingelheim Investigational Site, Hartha
  - Boehringer Ingelheim Investigational Site, Heidelberg
  - Boehringer Ingelheim Investigational Site, Heidenheim
  - Boehringer Ingelheim Investigational Site, Heilbronn
  - Boehringer Ingelheim Investigational Site, Hemmingen
  - Boehringer Ingelheim Investigational Site, Hildburghausen
  - Boehringer Ingelheim Investigational Site, Hildesheim
  - Boehringer Ingelheim Investigational Site, Homburg/Saar
  - Boehringer Ingelheim Investigational Site, Hoyerswerda
  - Boehringer Ingelheim Investigational Site, Ingolstadt
  - Boehringer Ingelheim Investigational Site, Kamen
  - Boehringer Ingelheim Investigational Site, Karlsruhe
  - Boehringer Ingelheim Investigational Site, Kaufbeuren
  - Boehringer Ingelheim Investigational Site, Kempten
  - Boehringer Ingelheim Investigational Site, Kiel
  - Boehringer Ingelheim Investigational Site, Koblenz
  - Boehringer Ingelheim Investigational Site, Köthen
  - Boehringer Ingelheim Investigational Site, Krefeld
  - Boehringer Ingelheim Investigational Site, Landshut
  - Boehringer Ingelheim Investigational Site, Langenhagen
  - Boehringer Ingelheim Investigational Site, Leipzig
  - Boehringer Ingelheim Investigational Site, Leonberg
  - Boehringer Ingelheim Investigational Site, Loerrach
  - Boehringer Ingelheim Investigational Site, Ludwigsburg
  - Boehringer Ingelheim Investigational Site, Lübeck
  - Boehringer Ingelheim Investigational Site, Lüdenscheid
  - Boehringer Ingelheim Investigational Site, Lüneburg
  - Boehringer Ingelheim Investigational Site, Magdeburg
  - Boehringer Ingelheim Investigational Site, Mainz
  - Johannes-Gutenberg-Universität Mainz, Mainz
  - Boehringer Ingelheim Investigational Site, Mannheim
  - Boehringer Ingelheim Investigational Site, Marburg
  - Boehringer Ingelheim Investigational Site, Markkleeberg
  - Boehringer Ingelheim Investigational Site, Minden
  - Boehringer Ingelheim Investigational Site, Mittweida
  - Boehringer Ingelheim Investigational Site, Moers
  - Boehringer Ingelheim Investigational Site, Mönchengladbach
  - Boehringer Ingelheim Investigational Site, Mühlhausen
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Münster
  - Boehringer Ingelheim Investigational Site, Neu-Isenburg
  - Boehringer Ingelheim Investigational Site, Neu-Ulm
  - Boehringer Ingelheim Investigational Site, Neubrandenburg
  - Boehringer Ingelheim Investigational Site, Neuss
  - Boehringer Ingelheim Investigational Site, Neuwied
  - Boehringer Ingelheim Investigational Site, Niesky
  - Boehringer Ingelheim Investigational Site, Nordhausen
  - Boehringer Ingelheim Investigational Site, Nortorf
  - Boehringer Ingelheim Investigational Site, Oschatz
  - Boehringer Ingelheim Investigational Site, Oschersleben
  - Boehringer Ingelheim Investigational Site, Papenburg
  - Boehringer Ingelheim Investigational Site, Potsdam
  - Boehringer Ingelheim Investigational Site, Rathenow
  - Boehringer Ingelheim Investigational Site, Recklinghausen
  - Boehringer Ingelheim Investigational Site, Regensburg
  - Boehringer Ingelheim Investigational Site, Rehau
  - Boehringer Ingelheim Investigational Site, Remscheid
  - Boehringer Ingelheim Investigational Site, Reutlingen
  - Boehringer Ingelheim Investigational Site, Rhaunen
  - Boehringer Ingelheim Investigational Site, Rostock
  - Boehringer Ingelheim Investigational Site, Rüdersdorf
  - Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site, Saarbrücken
  - Boehringer Ingelheim Investigational Site, Saarlouis
  - Boehringer Ingelheim Investigational Site, Saint Ingbert
  - Boehringer Ingelheim Investigational Site, Schrobenhausen
  - Boehringer Ingelheim Investigational Site, Schwabach
  - Boehringer Ingelheim Investigational Site, Schwäbisch Gmünd
  - Boehringer Ingelheim Investigational Site, Schweinfurt
  - Boehringer Ingelheim Investigational Site, Schwetzingen
  - Boehringer Ingelheim Investigational Site, Siegen
  - Boehringer Ingelheim Investigational Site, Simmern
  - Boehringer Ingelheim Investigational Site, Sindelfingen
  - Boehringer Ingelheim Investigational Site, Singen
  - Boehringer Ingelheim Investigational Site, Solingen
  - Boehringer Ingelheim Investigational Site, Sonneberg
  - Boehringer Ingelheim Investigational Site, Stade
  - Boehringer Ingelheim Investigational Site, Steinhagen
  - Boehringer Ingelheim Investigational Site, Stolberg
  - Boehringer Ingelheim Investigational Site, Stuttgart
  - Boehringer Ingelheim Investigational Site, Teuchern
  - Boehringer Ingelheim Investigational Site, Ulm
  - Boehringer Ingelheim Investigational Site, Uttenreuth
  - Boehringer Ingelheim Investigational Site, Vechta
  - Boehringer Ingelheim Investigational Site, Velbert
  - Boehringer Ingelheim Investigational Site, Verden an der Aller
  - Boehringer Ingelheim Investigational Site, Vöhringen
  - Boehringer Ingelheim Investigational Site, Waiblingen
  - Boehringer Ingelheim Investigational Site, Waren
  - Boehringer Ingelheim Investigational Site, Welzheim
  - Boehringer Ingelheim Investigational Site, Weyhe
  - Boehringer Ingelheim Investigational Site, Wiesbaden
  - Boehringer Ingelheim Investigational Site, Wiesloch
  - Boehringer Ingelheim Investigational Site, Witten
  - Boehringer Ingelheim Investigational Site, Wolfsburg
  - Boehringer Ingelheim Investigational Site, Wuppertal
  - Boehringer Ingelheim Investigational Site, Zerbst
  - Boehringer Ingelheim Investigational Site, Zwickau